CLINICAL TRIAL: NCT05680142
Title: Efficacy of Cervical Erector Spina Plane Block and Superficial Cervical Plexus Block in Anterior Cervical Disc and Fusion Surgery
Brief Title: Regional Analgesia for Anterior Cervical Disc and Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Ergün Mendeş, Specialist Doctor, Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Interventional; 2023.06.232 (Other: Basaksehir Cam and Sakura City Hospital)
Record Dates: First submitted 2022-11-22; First posted 2023-01-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain; Shoulder Pain; Anesthesia, Local; Disc Herniation
Keywords: cervical erector spinae block; anterior cervical disc and fusion surgery; postoperative analgesic consumption; superficial cervical plexus block
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain; Intervertebral Disc Displacement | interventions — small cardioactive peptide B

STUDY DESIGN:
Intervention Model Description: In the preoperative period, the participant groups will be divided into two separate groups, Group cESP and Group sCPB, according to the type of block applied.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: After the block, another anesthetist who did not know which group the patient belonged to was included in the study blindly. The patients were taken to the recovery unit in the postoperative period, and their analgesic needs, frequency of nausea and vomiting, VAS scores and additional problems were followed up by the nurse who was blindly included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group sCPB (Active Comparator): Superficial cervical plexus block, patients who applied sCPB for postoperative pain
  Interventions: Drug: superficial cervical plexus block
- Group cESP (Active Comparator): Cervical erector spinae plane block, patients who applied cervical ESP block for postoperative pain
  Interventions: Drug: cervical erector spinae plane block

INTERVENTIONS:
Drug: superficial cervical plexus block — The superficial cervical plexus block is applied as part of our routine protocol for postoperative pain control. Group sCPB will be administered from the C4 level by entering the posterior border of the sternocleidomastoid muscle from the right side of the neck.
  Other Names: sCPB
  Arms: Group sCPB
Drug: cervical erector spinae plane block — The cervical erector spinae plane block is applied as part of our routine protocol for postoperative pain control. Group cESP is applied to the fascia between the semispinalis capitis muscle and the posterior scalene muscle of the C6 or C7 transverse process.
  Other Names: cESP
  Arms: Group cESP

SUMMARY:
Erector Spina Plane (ESP) block has been widely used in recent years, and it is also used in the control of postoperative analgesia in many types of surgery due to its proximity to the central area and its wide spread feature. In this study, the investigators aimed to demonstrate the effectiveness of ESP block on postoperative pain management in anterior cervical disc and fusion surgeries.

DETAILED DESCRIPTION:
This study includes ASA I-II patients aged 18-65 years who will undergo Anterior Cervical Disc and Fusion Surgery at C5 or C6 level under general anesthesia under elective conditions. In the preoperative period, the participant groups will be divided into two separate groups, Group cESP and Group sCPB, according to the type of block applied.

Groups will be compared according to demographic data, duration of surgery, perioperative drug consumption, postoperative pain scores, additional analgesic requirement and presence of shoulder pain. The blocks will be applied with the help of an 8-12 mHz linear probe after the patients are determined by the closed envelope method. In group cESP, block will be applied using in-plane technique at the level of C6 or C7 transverse vertebral corpus in the fascia between the semispinalis capitis muscle and the posterior scalene muscle. During the block, a total of 20 mL volume of 0.25% bupivacaine concentration will be given bilaterally to all patients. Group sCPB will be administered using 10 mL of 0.25% bupivacaine by entering from the C4 level from the right side of the neck from the posterior side of the sternocleidomastoid muscle. It was planned to routinely administer 10 mg/kg paracetamol and 2x10 mg tenoxicam iv to all patients for postoperative pain control. Patients will be taken to the recovery unit in the postoperative period, where their analgesic needs, frequency of nausea-vomiting, VAS scores, and additional problems will be followed up by the nurse who was included in the study blindly. After 1 hour of follow-up in the Recovery Unit, the participants will be directed to the service. The participants' VAS scores and additional analgesic needs will be recorded at 6, 12, and 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) Classification I-II
* Anterior Cervical Disc and Fusion Surgery

Exclusion Criteria:

* Patients with bleeding diathesis
* Neurological disease,
* BMI (Body Mass Index) less than 19 or greater than 30
* The presence of infection in the neck area
* Patients who do not accept the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Qualitif of Recovery-15 (QoR-15) | Postoperative 24th hour
  The QoR-15 scale is a unidimensional measurement of quality of recovery measured in five domains: physical comfort, pain, physical independence, psychological support, and emotional state. The QoR-15 scale provides a score ranging from 0 to 150, with a high score indicating a good quality of recovery
VAS (Visual Analog Scala) score | Postoperative 24th hour
  The patients were followed up with a VAS score between 0-10 in the postoperative period. A VAS score of 0 was defined as no pain, and 10 as the most severe pain imaginable.

SECONDARY OUTCOMES:
Analgesic consumption | Postoperative 24th hour
  The value in mg of the amount of analgesic consumed in the postoperative period. It was administered with a PCA device that had regular infusions and was able to deliver bolus doses at regular intervals.
Postoperative nausea and vomiting | Postoperative 24th hour
  The frequency of nausea and vomiting in the postoperative period was calculated according to the Numeric Rank Score (NRS), which ranged from 0 to 3. Nausea-vomiting status of the patients: 0 points if there is no nausea and vomiting; 1 point if there is nausea, no vomiting; It is scored as 2 points if there is vomiting once and 3 points if there are two or more vomiting attacks.
Chronic Pain | 1 month after surgery
  Evaluation of shoulder pain level in terms of chronic pain in the postoperative period. It was evaluated using the VAS (Visual Analog Scala) score. The patients were followed up with a VAS score between 0-10 in the postoperative period. A VAS score of 0 was defined as no pain, and 10 as the most severe pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Ergun Mendes, Principal Investigator — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Ergun Mendes, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Elsharkawy H, Ince I, Hamadnalla H, Drake RL, Tsui BCH. Cervical erector spinae plane block: a cadaver study. Reg Anesth Pain Med. 2020 Jul;45(7):552-556. doi: 10.1136/rapm-2019-101154. Epub 2020 Apr 21. PMID 32321860
- [Background] Mariappan R, Mehta J, Massicotte E, Nagappa M, Manninen P, Venkatraghavan L. Effect of superficial cervical plexus block on postoperative quality of recovery after anterior cervical discectomy and fusion: a randomized controlled trial. Can J Anaesth. 2015 Aug;62(8):883-90. doi: 10.1007/s12630-015-0382-3. Epub 2015 Apr 14. PMID 25869024